CLINICAL TRIAL: NCT04990557
Title: CRISPR/Cas9-modified Human T Cell ( PD-1and ACE2 Knockout Engineered T Cells ) for Inducing Long-term Immunity in COVID-19 Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Ramadan mohamed Elkazzaz (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Ramadan mohamed Elkazzaz, Clinical Researcher, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Novel Treatment for Covid-19
Record Dates: First submitted 2021-08-01; First posted 2021-08-04 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A - Two cycles (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) and ACE2 gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1/ACE2 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients.
  A total of 1 x 10^7/kg PD-1and ACE2 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Interventions: Drug: PD-1 and ACE2 Knockout T Cells
- B- Two cycles (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) and ACE2 gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1/ACE2 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients.
  A total of 1 x 10^7/kg PD-1 and ACE2 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  A total of 2 x 10^7/kg PD-1and ACE2 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Interventions: Drug: PD-1 and ACE2 Knockout T Cells
- C- Two cycles (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) and ACE2 gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1/ACE2 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients.
  A total of 4 x 10^7/kg PD-1 and ACE2 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Interventions: Drug: PD-1 and ACE2 Knockout T Cells

INTERVENTIONS:
Drug: PD-1 and ACE2 Knockout T Cells — Autologous lymphocytes are collected and both PDCD1 and ACE2 gene knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment
  Arms: A - Two cycles
Drug: PD-1 and ACE2 Knockout T Cells — Autologous lymphocytes are collected and both PDCD1 and ACE2 gene knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment
  Arms: B- Two cycles
Drug: PD-1 and ACE2 Knockout T Cells — Autologous lymphocytes are collected and both PDCD1 and ACE2 gene knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment
  Arms: C- Two cycles

SUMMARY:
T-cell exhaustion may limit long-term immunity in COVID-19 patients. T cells can lose their ability to fight viruses and tumors when they have prolonged exposure to these enemies. New data suggests people who experience mild COVID-19 symptoms show the molecular signs of exhausted memory T cells and therefore could have a reduced ability to fight reinfection. On contrary people who develop severe COVID-19 symptoms may be better protected from reinfection. A recent study reported that the 82.1% of COVID-19 cases displayed low circulating lymphocyte counts . It has been reported that, in the case of chronic viruses, continuous PD-1 expression causes T-cell exhaustion, and impairs the ability of killing the infectious cells . The adumbration of patients with COVID-19 is characterized by a diminished lymphocyte percentage, with a similar proportion of CD4+ and CD8+ T-cells. The quantity of T-cells, mostly CD8+ T-cells, presenting high expression rates of late activity marker CD25 and exhaustion marker PD-1 increases. Therefore, SARS-CoV-2 is able to make changes by modifying the acquired immune system, including B and T cells. According to experiments, PD-1's expression, as an important factor in the induction and maintenance of circumferential tolerance keeping the stability of T-cells, has been found to have a higher percentage in different cells of COVID-19 patients. In an experiment conducted by Diao et al., on the patients with SARS-CoV-2, it was observed that the expression of PD-1 on the surface of T-cells was increased significantly; it was also shown that during the SARS-CoV-2 -induced disease, additional expressions of PD-1 and Tim-3 on the T-cells were directly related to the disease's severity; the factors that were also increased in other viral infections. T cell exhaustion" phenomenon could be reversed relatively easily, for example when the T cells are no longer exposed to the virus or tumor. But unfortunately, although exhausted T cells recovered from chronic infection (REC-TEX) regain some function and features of memory T cells (TMEM), they retain epigenetic scars indicating the control of gene expression is "locked in" to their exhaustion history. Once T cells become exhausted, they remain fundamentally 'wired' to be exhausted-thus it may be hard to get them to become effective virus- and cancer-fighters again," said John Wherry, PhD, chair of the department of Systems Pharmacology and Translational Therapeutics and director of the Penn Institute of Immunology in the Perelman School of Medicine at the University of Pennsylvania. Furthermore, COVID-19 may infect T lymphocyte cells and induce apoptosis and apoptotic markers. Lymphocytopenia was also found in the Middle East respiratory syndrome (MERS) cases. MERS-CoV can directly infect human primary T lymphocytes and induce T-cell apoptosis through extrinsic and intrinsic apoptosis pathways, but it cannot replicate in T lymphocytes. However, it is unclear whether SARS-CoV-2 can also infect T cells, resulting in lymphocytopenia. A study showed that T cells express a very low expression level of hACE2 on its cell surface and T-cell lines were significantly more sensitive to SARS-CoV-2 infection when compared with SARS-CoV . In other words, these results tell us that T lymphocytes may be more permissive to SARS-CoV-2 infection. Therefore, it is plausible that the S protein of SARS-CoV-2 might mediate potent infectivity, even on cells expressing low hACE2, which would, in turn, explain why the transmission rate of SARS-CoV-2 is so high. Through recent advances in genomic editing, T cells can now be successfully modified via CRISPR/Cas9 technology. For instance, engaging (post-)transcriptional mechanisms to enhance T cell cytokine production, the retargeting of T cell antigen specificity or rendering T cells refractive to inhibitory receptor signaling can augment T cell effector function. Therefore, CRISPR/Cas9-mediated genome editing might provide novel strategies for inducing long term immunity against COVID-19.Immunotherapies with autologous T cells have become a powerful treatment option for many diseases like viral infection or cancer. These include the adoptive isolation and transfer of naturally-occurring virus/tumor-specific T cells and the transfer of T lymphocytes that have been genetically modified . According to the investigator, exhausted virus-reactive CD8+ memory T cells will be isolated from patients with mild infection using a modified antigen-reactive T cell enrichment (ARTE) assay. exhausted virus-reactive CD8+ memory T cells will be collected and both Programmed cell death protein 1(PDCD1) gene and ACE2 gene will be knocked out by CRISPR Cas9 in the laboratory. The lymphocytes will be selected and expanded ex vivo and infused back into patients.

DETAILED DESCRIPTION:
This study will assess the safety of PD-1 and ACE2 knockout engineered T cells as genetically modified memory T cells capable of providing long-term immunity against COVID-19 by remembering and killing the virus if it is reintroduced. Blood samples will also be collected for research purposes. This is a dose-escalation study of ex-vivo knocked-out, expanded, and selected PD-1 and ACE2 knockout-T cells from autologous origin. Patients are assigned to 1 of 3 treatment groups to determine the maximal tolerant dose. After the lower number of cycles are considered tolerant, an arm of the next higher number of cycles will be open to next patients. Biomarkers and immunological markers are collected and analyzed as well. According to the investigator, exhausted virus-reactive CD8+ memory T cells will be isolated from patients with mild infection using a modified antigen-reactive T cell enrichment (ARTE) assay. exhausted virus-reactive CD8+ memory T cells will be collected and Programmed cell death protein 1(PDCD1) gene and ACE2 gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 and ACE2 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. A total of 2 x 10^7/kg PD-1 and ACE2 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who recently recovered from mild COVID-19 disease (First, second and third infection).
* Major organs function normally.
* Women at pregnant ages should be under contraception..
* Willing and able to provide informed consent

Exclusion Criteria

* Blood-borne infectious disease, e.g. hepatitis B.:
* History of mandatory custody because of psychosis or other psychological disease inappropriate for treatment deemed by treating physician.
* With other immune diseases, or chronic use of immunosuppressants or steroids.
* Compliance cannot be expected.
* Other conditions requiring exclusion deemed by physician

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events and/or Dose Limiting Toxicities as a Measure of Safety and Tolerability of Dose of PD-1 Knockout T Cells Using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in Patients | Dose Escalation - Approximately 5 months

SECONDARY OUTCOMES:
Number of Patients With Overall Response to the reinfection | 10 months
All cause mortality rate | Measured from Day 0 through Day 180
  The time from the date of first edited T cell infusion to the date of reinfection with COVID-19 or death due to any reason.
Proportion of patients with upregulated inflammatory factors | 1 month and 3 month
  Upregulated inflammatory factors will be measured at different timepoint
Serum levels of IL-6,TNF,TLR3,CRP, ESR and Type I interferon | 1 month and 3 month
  Serum levels of IL-6,TNF,TLR3,CRP, ESR and Type I interferon will be measured at different timepoint
Absolute lymphocyte counts (CD4,CD8 and CD25+FOXP3+ Regulatory T) | 1 month and 3 month
  Absolute lymphocyte counts (CD4,CD8 and CD25+FOXP3+ Regulatory T) will be measured at different timepoint
Safety-Hematology | Measured from Day 0 through Day 180
  white blood cells (WBC) Differential cell counts should be performed at baseline, at each visit during PD-1 Knockout Engineered T Cells infusion phase and thereafter at investigators discretion. Clinical status and laboratory parameters are to be followed using individual institutional guidelines and the best clinical judgment of the responsible physician, which can involve more frequent testing.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud R Elkazzaz, M.Sc of Biochemistry, Principal Investigator — Faculty of science Damietta university